CLINICAL TRIAL: NCT00964613
Title: Pars Plana Surgical Capsulotomy for Posterior Capsular Opacification
Acronym: Capsulotomy
Status: Completed | Type: Observational
Sponsor: Dow University of Health Sciences (Other)
Collaborators: Pakistan Ministry of Health (Other Government)
Responsible Party: Principal Investigator, Jamshed Ahmed, Assistant Professor, Dow University of Health Sciences
Other Study IDs: Surgical Capsulotomy
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Blindness
Keywords: Pars Plana; Surgical Capsulotomy; Posterior capsule opacification; visual outcome; Complications
MeSH Terms: conditions — Blindness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Cataract is a leading cause of Global blindness. After cataract surgery nearly half of the people become blind due to posterior capsular opacification. The only solution for this problem is LASER capsulotomy. Laser machine is not available in remote areas especially in underdeveloped countries. The solution of this problem is surgical capsulotomy which can be performed any where.

DETAILED DESCRIPTION:
posterior capsular opacification is treated by YAG laser capsulotomy. this require sophisticated technology ans specific environment which is not possible in underdeveloped countries. we describe a method in which posterior capsular opacification could be managed by using only a 27 Gauge needle through pars plana. opacified posterior capsule is under tension that is why a small puncture results in a large central opening

ELIGIBILITY:
Inclusion Criteria:

* Patients with Posterior capsular opacification
* Both Sexes
* All ages

Exclusion Criteria:

* Retinal disease
* Uncontrolled Glaucoma
* Corneal opacity

Ages: 1 Year to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients having posterior capsular opacification
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)